CLINICAL TRIAL: NCT03827005
Title: The Acute Effects of L-arginine Supplementation on Flow-mediated Dilation After Resistance Exercise to Fatigue
Brief Title: L-arginine Supplementation and Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Principal Investigator, Kyle Hackney, Assistant Professor, North Dakota State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HE16235
Record Dates: First submitted 2018-07-01; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Healthy Adult
Keywords: L-arginine; flow mediated dilation; resistance exercise
MeSH Terms: interventions — Arginine; Starch

STUDY DESIGN:
Intervention Model Description: double blind, placebo, controlled -cross over
Who Masked: Participant, Investigator
Masking Description: blinding performed by co-investigator not involved with data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): 3 grams cornstarch once per day for one day.
  Interventions: Dietary Supplement: L-arginine; Dietary Supplement: Placebo
- L-arginine (Experimental): 3 g L-arginine once per day for one day.
  Interventions: Dietary Supplement: L-arginine; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-arginine — NOW Foods, Bloomingdale, IL
Dietary Supplement: Placebo — InHealth Specialty Pharmacy, Fargo, ND
  Other Names: cornstarch

SUMMARY:
The purpose of this study was to examine the acute endothelial, cardiovascular, and performance responses to L-arginine by assessing flow-mediated dilation (FMD) and heart rate variability (HRV) both before and after resistance exercise to fatigue. Thirty (15 male, 15 female) physically active participants volunteered for a randomized, cross-over, double-blind, placebo- controlled clinical trial. Participants completed five sets of elbow extension-flexion exercise after consumption of either 3 g of placebo or 3 g L-arginine.

DETAILED DESCRIPTION:
Participants Thirty healthy, physically active males (n=15) and females (n=15), 18-25 years of age completed the study. Subjects had not participated in another clinical trial or consumed another study related investigation product within 30 days of enrollment. If a supplement containing L-arginine or other nitrate precursors was being taken, a three-week washout period was conducted before participation. All procedures were approved in advance by the North Dakota State University Institutional Review Board and written consent was obtained.

Protocol A randomized, double-blind, placebo-controlled research design was implemented for this investigation. Prior to the randomized testing sessions, participants completed a anthropometric measurements and familiarization session which included:: collection of participant age, height (Seca 213, Chino, CA), and body mass data (Detecto, Webb City, MO) and familiarization with the Biodex Dynamometer (Biodex Medical Systems, Shirley, NY), ultrasound (Philips Ultrasound, Bothell, WA), and electronic sphygmomanometer (Hokanson Rapid Cuff Inflation System, Bellevue, WA) procedures. Participants then reported to the laboratory for two testing sessions, each separated by at least a 48 hours washout period. Testing sessions were conducted at the same time of day to account for circadian variation. Participants entered the trial sessions on an 8-our fast, but were encouraged to arrive at the session well-hydrated. The participants were instructed not to exercise or consume caffeine 24 hours prior to trial time or use toothpaste, chewing gum, or mouthwash the morning of the trials, due to the possible effects on nitric oxide absorption. All females tested negative for pregnancy based on a urinary pregnancy test (Clinical Guard, Atlanta, GA) prior to each trial session. At the start of the trial, participants rested for 5 minutes while sitting.

Endothelial responses were measured by a technique termed flow mediated vasodilation (FMD) which assessed the maximal vasodilatory response to shear stress. FMD was measured in accordance with recommendations from the International Brachial Artery Reactivity Task Force. A Philips HD11XE ultrasound system (Philips, Amsterdam, NL) equipped with 2D imaging, color and spectral Doppler, and a high-frequency vascular transducer was used for the protocol. The participants laid supine with the right arm inside a pillow for a stabilizer. Probe placement was on the brachial artery, above the antecubital fossa in the longitudinal place. Continuous 2D imaging was used to take an initial brachial artery diameter for 10 seconds to determine the resting artery diameter (to cover the full cardiac cycle). Probe placement was outlined with a marker. A Hokanson E20 electronic sphygmomanometric cuff and rapid cuff inflation system (Bellevue, WA) was placed on the middle of the forearm and inflated to 50 mmHg above systolic blood pressure for five mins and cuff placement was marked with a marker. Upon release of the cuff, the ultrasound probe was placed in the same area in which the first measure was taken. A continuous 2D imaging was used from cuff release to 120 seconds post-release. The average of three diameters measured using RadiAnt DICOM software was used for determination of FMD (%), which was expressed as the change in post-stimulus diameter as a percentage of baseline diameter.

Measures of the cardiovascular system included heart rate variability (HRV). HRV were recorded using a Polar H7 Bluetooth strap (Polar, Bethpage, NY) combined Personal Pro Elite HRV smartphone application (elitehrv.com) over 5 min intervals then further analyzed with Kubios software using the "very low" artifact correction setting. HRV explored the differences in beat-to-beat intervals based on the time (milliseconds) between adjacent R to R (RR) peaks within a PQRST waveform. HRV provides a dynamic, sensitive meter of the balance or tone between the two branches of the autonomic nervous system, sympathetic (SNS) and parasympathetic (PNS), RMSSD and pNN50 are also the most commonly used HRV measures and were used in this study.

After baseline measurements were collected, the participants consumed either 6 capsules (3 g) of L-arginine (NOW Foods, Bloomingdale, IL) or 6 capsules of corn starch, placebo (3 g) which had an identical appearance (InHealth Specialty Pharmacy, Fargo, ND). Each supplement was consumed with 12 oz. of water. The participant then rested for 55 minutes to ensure enough time for digestion, absorption and availability. At 55 minutes post-supplementation, participants completed a 5 minutes warm up using a cycle ergometer (Monark 828E, Vansbro, SV). Sixty minutes post-supplementation, participants completed elbow flexion and extension exercise with their right arm on an isokinetic dynamometer to determine the elbow flexor and extensor peak torque.The exercise protocol, designed to induce fatigue, consisted of five sets of 10 maximal isokinetic extension repetitions of the elbow joint at 90º per second with 30 seconds of rest in between sets. Participants were instructed and encouraged to use full-force for all sets. Isometric peak torque was measured prior to and thirty seconds after exercise to determine the fatigue percentage. Dynamometer settings remained constant for each testing session as recorded during the anthropometric and familiarization session. At 10 minutes post-exercise, which was 120 minutes after supplement consumption, FMD and HRV were measured for the final time.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* physically active

Exclusion Criteria:

* previous clinical trial
* pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self reported
Enrollment: 30 (Actual)
Dates: Start 2016-07-16 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Flow mediated dilation 120 seconds post-cuff release | Change from Baseline and 120 seconds
  Flow mediated dilation was measured using a A Philips HD11XE ultrasound system (Philips, Amsterdam, NL) equipped with 2D imaging, color and spectral Doppler, and a high-frequency vascular transducer.
Change in Heart Rate Variability 10 minutes after intervention | Change from Baseline and 10 minutes post-exercise
  Hear rate variability was recorded using a Polar H7 Bluetooth strap (Polar, Bethpage, NY) combined Personal Pro Elite HRV smartphone application (elitehrv.com) over 5 minutes intervals then further analyzed with Kubios software

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvares TS, Conte CA, Paschoalin VM, Silva JT, Meirelles Cde M, Bhambhani YN, Gomes PS. Acute l-arginine supplementation increases muscle blood volume but not strength performance. Appl Physiol Nutr Metab. 2012 Feb;37(1):115-26. doi: 10.1139/h11-144. Epub 2012 Jan 17. PMID 22251130
- [Background] Alvares TS, Meirelles CM, Bhambhani YN, Paschoalin VM, Gomes PS. L-Arginine as a potential ergogenic aid in healthy subjects. Sports Med. 2011 Mar 1;41(3):233-48. doi: 10.2165/11538590-000000000-00000. PMID 21395365
- [Background] Bondonno CP, Croft KD, Hodgson JM. Dietary Nitrate, Nitric Oxide, and Cardiovascular Health. Crit Rev Food Sci Nutr. 2016 Sep 9;56(12):2036-52. doi: 10.1080/10408398.2013.811212. PMID 25976309
- [Background] Bai Y, Sun L, Yang T, Sun K, Chen J, Hui R. Increase in fasting vascular endothelial function after short-term oral L-arginine is effective when baseline flow-mediated dilation is low: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2009 Jan;89(1):77-84. doi: 10.3945/ajcn.2008.26544. Epub 2008 Dec 3. PMID 19056561
- [Background] Kapadia MR, Eng JW, Jiang Q, Stoyanovsky DA, Kibbe MR. Nitric oxide regulates the 26S proteasome in vascular smooth muscle cells. Nitric Oxide. 2009 Jun;20(4):279-88. doi: 10.1016/j.niox.2009.02.005. Epub 2009 Feb 20. PMID 19233305
- [Background] Arnal JF, Dinh-Xuan AT, Pueyo M, Darblade B, Rami J. Endothelium-derived nitric oxide and vascular physiology and pathology. Cell Mol Life Sci. 1999 Jul;55(8-9):1078-87. doi: 10.1007/s000180050358. PMID 10442089
- [Background] Fahs CA, Heffernan KS, Fernhall B. Hemodynamic and vascular response to resistance exercise with L-arginine. Med Sci Sports Exerc. 2009 Apr;41(4):773-9. doi: 10.1249/MSS.0b013e3181909d9d. PMID 19276857